CLINICAL TRIAL: NCT05264506
Title: A Phase 3, Open-label, Multi-center, Single-arm Study to Assess Contraceptive Efficacy and Safety of the Nomegestrol Acetate + 17β-estradiol Combined Oral Contraceptive (OG-8175A) in Premenopausal Females Aged 14 to 35 Years (Inclusive)
Brief Title: Contraceptive Efficacy and Safety of NOMAC-E2 Combined Oral Contraceptive
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision to stop the study early and complete all required study close-out activities. This decision was made for business reasons unrelated to safety. None of the pre-specified efficacy endpoints were analyzed.
Sponsor: Organon and Co (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OG-8175A-023
Record Dates: First submitted 2022-01-28; First posted 2022-03-03 (Actual); Results first posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-09

CONDITIONS: Contraception
Keywords: Birth control methods; Contraceptive; Postmenarcheal Premenopausal Women; Hormonal; Sexually Active
MeSH Terms: interventions — nomegestrol acetate; Estradiol

STUDY DESIGN:
Intervention Model Description: Single Arm Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nomegestrol Acetate + 17β-estradiol (NOMAC-E2; OG-8175A) (Experimental): The NOMAC-E2 COC active tablets contain 2.5 mg NOMAC and 1.5 mg E2 and will be used in a 24/4 regimen, i.e., 28-day cycles with 24 days of active tablet intake followed by 4 days of placebo tablet intake.
  Interventions: Drug: NOMAC-E2 COC

INTERVENTIONS:
Drug: NOMAC-E2 COC — Dosage Formulation: Film-coated Tablet Unit Dose Strength: Nomegestrol acetate (NOMAC) 2.5 mg and estradiol (E2) 1.5 mg; Each blister strip contains 28 tablets: 24 tablets with the active drug (number 1 to 24) and 4 tablets with placebo (number 25 to 28).
  Dosing Instructions: oral. Take 1 tablet daily at about the same time as directed.
  Other Names: Nomegestrol acetate / estradiol

SUMMARY:
The purpose of this study is evaluating Contraceptive Efficacy and Safety of NOMAC-E2 Combined Oral Contraceptive in Premenopausal Females Aged 14 to 35 Years (Inclusive).

DETAILED DESCRIPTION:
This is a Phase 3, Open-label, Multi-center, Single-arm Study to Assess Contraceptive Efficacy and Safety of the Nomegestrol Acetate + 17β-estradiol Combined Oral Contraceptive (OG-8175A) in Premenopausal Females Aged 14 to 35 Years (Inclusive). Potential participants must be sexually active and engage in heterosexual vaginal intercourse at least once per month with a partner who is not known to be subfertile, sterilized, or infertile, and should not routinely use any other form of contraception.

A total of 2,680 fertile premenopausal women aged 14 to 35 years (inclusive) will be screened to achieve about 1,878 (with at least 657 participants with BMI ≥30 kg/m2) being allocated to study treatment. Over 1,000 total participants are expected to complete 1 year of treatment (13 cycles).

The total duration of study participation will be up to 60 weeks, which includes a Pre-treatment Period of approximately 6 weeks, a Treatment Period of 52 weeks, and a Follow-up Period of 2 weeks after the last intake of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Postmenarcheal, premenopausal female aged 14 to 35 years (inclusive)
* At risk for pregnancy (including heterosexual vaginal intercourse at least once a month and not sterilized).
* No desire for pregnancy within 1 year following screening and is not intending to use any other form of contraception
* Good physical and mental health
* History of regular menstrual cycles prior to the use of any hormonal contraceptive.
* Able and willing to adhere study procedures

Exclusion Criteria:

* Current known or expected pregnancy
* History of subfertility or infertility
* Less than 2 normal menstrual cycles following recent pregnancy of gestational age
* Breastfeeding within 2 months of study drug start
* Known HIV infection
* Untreated gonorrhea, chlamydia, or trichomonas
* abnormal PAP within timeline of standard of care guidelines
* Unexplained/unresolved abnormal vaginal bleeding
* Presence/history of VTE, ATE, transient ischemic attack, angina pectoris, or claudication
* Higher risk for VTE
* Uncontrolled or severe hypertension
* Severe dyslipoproteinemia
* History of migraine with aura or focal neurological symptoms
* Diabetes mellitus (with either end-organ involvement or >20 years duration)
* Multiple cardiovascular risk factors
* History of pancreatitis associated with severe hypertriglyceridemia
* Presence/history of clinically significant liver disease
* History of malabsorptive surgical procedures
* History of malignancy in last 5 years
* Presence/history of meningioma
* Disease that may worsen under hormonal treatment
* Presence/history of severe depression (unless currently stable and asymptomatic)
* Known allergy/sensitivity to NOMAC-E2
* Drug or alcohol abuse/dependence in last 2 years
* Clinically relevant abnormal lab result at screening
* Expected use of other contraceptive medications or medications that induce liver enzymes during study
* Used another investigational drug within 2 months of study drug start

Ages: 14 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3055 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-01-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (102):
- United States (102):
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - SEC Clinical Research, Dothan, Alabama
  - Alliance for Multispecialty Research, LLC, Mobile, Alabama
  - Velocity Clinical Research, Mobile, Alabama
  - Mesa Obstetricians and Gynecologists, Mesa, Arizona
  - Desert Clinical Research, LLC/CCT Research, Mesa, Arizona
  - Velocity Clinical Research - Phoenix, Phoenix, Arizona
  - Precision Trials AZ, LLC, Phoenix, Arizona
  - Alliance for Multispecialty Research, Tempe, Arizona
  - Noble Clinical Research, Tucson, Arizona
  - Eclipse Clinical Research, Tucson, Arizona
  - Gardens Medical Center / Alliance Research Institute, Bell Gardens, California
  - Alliance Research Institute, LLC, Canoga Park, California
  - Advanced Investigative Medicine, Inc, Hawthorne, California
  - Marvel Clinical Research, Huntington Beach, California
  - Om Research LLC, Lancaster, California
  - Empire Clinical Research, Pomona, California
  - WR-Women's Health Care Research, LLC, San Diego, California
  - WR-Medical Center For Clinical Research - San Diego, San Diego, California
  - Velocity Clinical Research, Denver, Colorado
  - Physicians' Research Options / Red Rocks OB/GYN, Lakewood, Colorado
  - CMR of Greater New Haven, LLC, Hamden, Connecticut
  - Alliance for Multispecialty Research, LLC, Coral Gables, Florida
  - Universal Axon Clinical Research, LLC, Doral, Florida
  - Alliance for Multispecialty Research, LLC, Fort Myers, Florida
  - Altus Research, Inc., Lake Worth, Florida
  - Accel Research Sites - St. Petersburg Clinical Research Unit, Largo, Florida
  - OB-GYN Associates of Mid-Florida, PA, Leesburg, Florida
  - Avantis Clinical Research, LLC, Miami, Florida
  - Miami Clinical Research, Miami, Florida
  - Admed Research, LLC, Miami, Florida
  - Genoma Research Group, Inc., Miami, Florida
  - Spotlight Research Center, LLC, Miami, Florida
  - New Age Medical Research Corporation, Miami, Florida
  - Quantum Clinical Trials, Miami Beach, Florida
  - Quality Research of South Florida, Miami Lakes, Florida
  - Healthcare Clinical Data, Inc., North Miami, Florida
  - Sensible Healthcare LLC, Ocoee, Florida
  - Innovation Medical Research Center, Palmetto Bay, Florida
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - R & B Medical Center LLC, Tampa, Florida
  - Comprehensive Clinical Research, LLC, West Palm Beach, Florida
  - Agile Clinical Research Trials, LLC, Atlanta, Georgia
  - Infinite Clinical Trials, Morrow, Georgia
  - Javara Inc / Privia Medical Group Georgia, LLC, Pooler, Georgia
  - WR-Mount Vernon Clinical Research, LLC, Sandy Springs, Georgia
  - Leavitt Clinical Research, Idaho Falls, Idaho
  - Women's Healthcare Associates P.A., Idaho Falls, Idaho
  - The Iowa Clinic, Ankeny, Iowa
  - Alliance for Multispecialty Research, LLC, El Dorado, Kansas
  - Alliance for Multispecialty Research, LLC, Newton, Kansas
  - Alliance for Multispecialty Research, LLC, Wichita, Kansas
  - Alliance for Multispecialty Research, LLC - Lexington, Lexington, Kentucky
  - Velocity Clinical Research - Covington, Covington, Louisiana
  - Velocity Clinical Research, Lafayette, Louisiana
  - Southern Clinical Research Associates, Metairie, Louisiana
  - Velocity Clinical Research, Metairie, Louisiana
  - Alliance for Multispecialty Research, LLC, New Orleans, Louisiana
  - Velocity Clinical Research, Slidell, Louisiana
  - Continental Clinical Solutions, Towson, Maryland
  - NECCR PrimaCare Research, LLC, Fall River, Massachusetts
  - Exordia Medical Research, Inc, Fall River, Massachusetts
  - Velocity Clinical Research, Gulfport, Mississippi
  - Alliance for Multispecialty Research, LLC, Kansas City, Missouri
  - Velocity Clinical Research, Grand Island, Nebraska
  - Velocity Clinical Research, Hastings, Nebraska
  - Velocity Clinical Research, Omaha, Nebraska
  - Jubilee Clinical Research, Inc, Las Vegas, Nevada
  - Essential Women's Health Associates, Las Vegas, Nevada
  - Alliance for Multispecialty Research, LLC, Las Vegas, Nevada
  - Planned Parenthood of Northern, Central, and Southern New Jersey, Perth Amboy, New Jersey
  - Albuquerque Clinical Trials, Inc, Albuquerque, New Mexico
  - Bosque Women's Care, Albuquerque, New Mexico
  - Meridian Clinical Research, LLC, Vestal, New York
  - Carolina Women's Research and Wellness Center, Durham, North Carolina
  - Carolina Institute For Clinical Research, Fayetteville, North Carolina
  - M3 Wake Research, Inc, Raleigh, North Carolina
  - University of Cincinnati Physicians, Cincinnati, Ohio
  - OB/GYN Associates of Erie, Erie, Pennsylvania
  - Clinical Research of Philadelphia, LLC, Philadelphia, Pennsylvania
  - Venus Gynecology, LLC, Myrtle Beach, South Carolina
  - Chattanooga Medical Research, LLC, Chattanooga, Tennessee
  - Alliance for Multispecialty Research, LLC, Knoxville, Tennessee
  - New Phase Research & Development, Knoxville, Tennessee
  - WR-Medical Research Center of Memphis, Memphis, Tennessee
  - Tekton Research, Inc, Austin, Texas
  - Helios Clinical Research, Burleson, Texas
  - Cedar Health Research, Dallas, Texas
  - Helios Clinical Research, Fort Worth, Texas
  - Javara Inc, Houston, Texas
  - Accurate Clinical Research, Inc, Houston, Texas
  - Clinical Trial Network, Houston, Texas
  - Texas Health Care, PLLC d/b/d Privia Medical Group - North Texas, Rowlett, Texas
  - Tekton Research, Inc, San Antonio, Texas
  - Javara Research, Stephenville, Texas
  - Javara Inc, Sugar Land, Texas
  - Helios Clinical Research - Weatherford, Weatherford, Texas
  - Wasatch Clinical Research, Salt Lake City, Utah
  - Javara Research, Forest, Virginia
  - Alliance for Multispecialty Research, LLC, Norfolk, Virginia
  - Tidewater Clinical Research, Norfolk, Virginia
  - Seattle Clinical Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 3,055 participants were screened for the study. Out of these 1,135 participants failed the screening process. One participant was found pregnant before starting treatment, however not identified as a screen failure
Period: Overall Study
Arm/Group | Nomegestrol Acetate + 17β-estradiol (NOMAC-E2; OG-8175A)
Started | 1919
Completed | 402
Not Completed | 1517
Not completed — Adverse Event | 59
Not completed — Lost to Follow-up | 204
Not completed — Protocol Violation | 185
Not completed — Pregnancy | 60
Not completed — Physician Decision | 6
Not completed — Non-compliance with Study Drug | 29
Not completed — Study termination | 677
Not completed — Withdrawal by Subject | 208
Not completed — Discontinued prior treatment | 89

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set consists of all participants who took at least one dose of the study treatment.
Groups:
- Nomegestrol Acetate + 17β-estradiol (NOMAC-E2; OG-8175A): The NOMAC-E2 COC active tablets contain 2.5 mg NOMAC and 1.5 mg E2 and will be used in a 24/4 regimen, i.e., 28-day cycles with 24 days of active tablet intake followed by 4 days of placebo tablet intake.
  NOMAC-E2 COC: Dosage Formulation: Film-coated Tablet Unit Dose Strength: Nomegestrol acetate (NOMAC) 2.5 mg and estradiol (E2) 1.5 mg; Each blister strip contains 28 tablets: 24 tablets with the active drug (number 1 to 24) and 4 tablets with placebo (number 25 to 28).
  Dosing Instructions: oral. Take 1 tablet daily at about the same time as directed.
Arm/Group | Nomegestrol Acetate + 17β-estradiol (NOMAC-E2; OG-8175A)
Number analyzed (Participants) | 1830
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.2 (4.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1830
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1004
  Not Hispanic or Latino | 817
  Unknown or Not Reported | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 15
  Asian | 29
  Native Hawaiian or Other Pacific Islander | 6
  Black or African American | 356
  White | 1358
  More than one race | 34
  Unknown or Not Reported | 32
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1830

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With On-treatment Pregnancies
Description: Raw count of the number of pregnancies that occurred while participants were taking study drug
Time Frame: 1 year
Population: All Participants as Treated Population, which consisted of all participants who took at least one dose of trial medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Nomegestrol Acetate + 17β-estradiol (NOMAC-E2; OG-8175A)
Number analyzed (Participants) | 1830
Participants | 57

2. Secondary Outcome: Proportion of Participants With an Adverse Event (Regardless on Potential Relationship to Study Drug)
Time Frame: 1 year
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Nomegestrol Acetate + 17β-estradiol (NOMAC-E2; OG-8175A)
Number analyzed (Participants) | 1830
participants | 485

3. Secondary Outcome: Proportion of Participants Who Prematurely Discontinue Study Drug Treatment
Time Frame: 1 year
Population: All Participants as Treated Population, which consisted of all randomized participants who took at least one dose of trial medication.
Measure: Number; unit: participants
Arm/Group | Nomegestrol Acetate + 17β-estradiol (NOMAC-E2; OG-8175A)
Number analyzed (Participants) | 1830
participants | 62

4. Secondary Outcome: Percentage of Participants With On-treatment Pregnancies With at Least One Completed Cycle
Description: Number of participants with on-treatment pregnancies as a percentage of the number of participants with at least one completed cycle
Time Frame: 1 year
Population: Participants with at least one completed cycle
Measure: Number; unit: percentage of participants
Arm/Group | Nomegestrol Acetate + 17β-estradiol (NOMAC-E2; OG-8175A)
Number analyzed (Participants) | 1756
percentage of participants | 3.1

5. Secondary Outcome: Number of Cycles of Exposure Prior to Pregnancy
Description: In participants who experienced on-treatment pregnancy, the mean number of completed treatment cycles prior to occurrence of the pregnancy (for participants with known date of conception)
Time Frame: 1 year
Population: Participants with a known date of conception
Measure: Mean (Standard Deviation); unit: completed cycles
Arm/Group | Nomegestrol Acetate + 17β-estradiol (NOMAC-E2; OG-8175A)
Number analyzed (Participants) | 31
completed cycles | 4.2 (3.47)

6. Secondary Outcome: Number of Participants With a Pregnancy, Based on Baseline BMI Categories (<30 kg/m2, ≥30 kg/m2)
Description: Raw count of the number of pregnancies that occurred while participants were taking study drug in each BMI category
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Nomegestrol Acetate + 17β-estradiol (NOMAC-E2; OG-8175A)
Number analyzed (Participants) | 57
Participants
  BMI <30 kg/m2 | 39
  BMI >=30 kg/m2 | 18

7. Secondary Outcome: Proportion of Participants With Bleeding-spotting Days
Description: Number of participants with bleeding-spotting days as a proportion of the number of participants who had at least one completed cycle
Time Frame: 28-day cycles across one year
Population: Participants with at least one completed cycle
Measure: Number; unit: participants
Arm/Group | Nomegestrol Acetate + 17β-estradiol (NOMAC-E2; OG-8175A)
Number analyzed (Participants) | 1756
participants | 1721

8. Secondary Outcome: Mean Number of Bleeding and/or Spotting Days Per Cycle
Description: For participants who had at least one completed cycle, the mean number of bleeding-spotting days per cycle
Time Frame: 28-day cycles across one year
Population: Participants with at least one completed cycle
Measure: Mean (Standard Deviation); unit: bleeding-spotting days
Arm/Group | Nomegestrol Acetate + 17β-estradiol (NOMAC-E2; OG-8175A)
Number analyzed (Participants) | 1756
bleeding-spotting days | 4.0 (3.44)

9. Secondary Outcome: Average Number of Bleeding-spotting Days Per Reference Period
Description: For participants with at least one completed reference period, the average number of bleeding-spotting days per reference period
Time Frame: 91-day reference periods across one year
Population: Participants with at least one completed reference period
Measure: Mean (Standard Deviation); unit: bleeding-spotting days
Arm/Group | Nomegestrol Acetate + 17β-estradiol (NOMAC-E2; OG-8175A)
Number analyzed (Participants) | 1518
bleeding-spotting days | 13.1 (8.54)

10. Secondary Outcome: Proportion of Participants With 8 or More Bleeding-spotting Days
Description: Proportion of participants who had at least one completed cycle with 8 or more bleeding-spotting days in a cycle
Time Frame: 28-day cycles across one year
Population: Participants with at least one completed cycle
Measure: Number; unit: participants
Arm/Group | Nomegestrol Acetate + 17β-estradiol (NOMAC-E2; OG-8175A)
Number analyzed (Participants) | 1756
participants | 709

11. Secondary Outcome: Mean NOMAC Concentration, Visit 3 Pre-Dose
Description: NOMAC concentrations assessed through use of sparse sampling
Time Frame: Treatment Week 5
Population: PK participants who completed Visit 3 pre-dose sampling
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Nomegestrol Acetate + 17β-estradiol (NOMAC-E2; OG-8175A)
Number analyzed (Participants) | 222
ng/mL | 32.26 (310.457)

12. Secondary Outcome: Mean NOMAC Concentration, Visit 3 Post-Dose
Description: NOMAC concentrations assessed through use of sparse sampling
Time Frame: Treatment Week 5
Population: PK participants who completed Visit 3 post-dose sampling
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Nomegestrol Acetate + 17β-estradiol (NOMAC-E2; OG-8175A)
Number analyzed (Participants) | 223
ng/mL | 73.61 (742.410)

13. Secondary Outcome: Mean NOMAC Concentration, Visit 4 Pre-Dose
Description: NOMAC concentrations assessed through use of sparse sampling
Time Frame: Treatment Week 17
Population: PK participants who completed Visit 4 pre-dose sampling
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Nomegestrol Acetate + 17β-estradiol (NOMAC-E2; OG-8175A)
Number analyzed (Participants) | 161
ng/mL | 36.01 (229.607)

14. Secondary Outcome: Mean NOMAC Concentration, Visit 4 Post-Dose
Description: NOMAC concentrations assessed through use of sparse sampling
Time Frame: Treatment Week 17
Population: PK participants who completed Visit 4 post-dose sampling
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Nomegestrol Acetate + 17β-estradiol (NOMAC-E2; OG-8175A)
Number analyzed (Participants) | 164
ng/mL | 58.01 (363.400)

ADVERSE EVENTS:
Time Frame: All AEs and SAEs were collected from the time of screening through the end of study/end of treatment visit, which was 14 to 19 days after the last intake of study drug, up to approximately 1 year, 1 month.
Description: The Safety Analysis Set consists of all participants who took at least one dose of the study treatment.
Arm/Group | Nomegestrol Acetate + 17β-estradiol (NOMAC-E2; OG-8175A)
All-Cause Mortality (participants affected / at risk) | 0/1830
Serious Adverse Events (participants affected / at risk) | 10/1830
Other Adverse Events (participants affected / at risk) | 0/1830
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nomegestrol Acetate + 17β-estradiol (NOMAC-E2; OG-8175A) (N=1830)
Burns third degree (Injury, poisoning and procedural complications) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 2 (2)
Bipolar disorder (Psychiatric disorders) | 1 (1)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 3 (3)

LIMITATIONS AND CAVEATS:
Due to the study's early discontinuation (for business reasons), a small number of participants completed the study prior to its discontinuation, limiting the data available for efficacy outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-08-30): https://cdn.clinicaltrials.gov/large-docs/06/NCT05264506/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-23): https://cdn.clinicaltrials.gov/large-docs/06/NCT05264506/SAP_002.pdf